CLINICAL TRIAL: NCT02388139
Title: Cardiovascular, Renal and Metabolic Profile in Patients With Acute Myocardial Infarction (AMI) Included in the Romanian National Programme of Primary Percutaneous Revascularisation - a Single Center Observational Study
Brief Title: Cardiovascular, Renal and Metabolic Profile in Patients With Acute Myocardial Infarction (REN-ACS)
Acronym: REN-ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, Professor coordinator, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: REN-ACS
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension, Renovascular; Renal Artery Stenosis; Myocardial Infarction
Keywords: acute myocardial infarction; renal artery stenosis
MeSH Terms: conditions — Hypertension, Renovascular; Renal Artery Obstruction; Myocardial Infarction | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum creatinine, serum urea, lipid profile, glycemia, haemoglobin, etc
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: renal artery angiography — preprocedural renal arteriogram is obtained after sterile preparation and draping of the patient, conscious sedation, infiltration of local anesthetic (lidocaine solution) at the femoral access site, placement of an arterial sheath in the femoral artery, and advancement of the renal guide catheter over a 0.035-in guidewire under fluoroscopic guidance. After the tip of the guide catheter is positioned at the ostium of the renal artery, an angiogram is obtained. After the guidewire is removed, the proximal end of the catheter is connected to a manifold, and 4-8 mL of contrast is manually injected during cineangiographic recording. An intravenous antithrombotic agent, usually heparin, is administered before the clinician proceeds with angioplasty.
Procedure: coronarography
Procedure: coronary angioplasty
  Other Names: pPCI
Procedure: pulse wave velocity measurement — is a measure of arterial stiffness with Sphigmocore device.
  Other Names: PWV
Procedure: body composition monitoring — using Fresenius device
  Other Names: BCM

SUMMARY:
Aims

* assessment of renal artery stenosis incidence in consecutive AMI patients included in the Romanian National Programme of Primary Percutaneous Revascularisation;
* generating a cardio-renal-metabolic profile in patients with renal atherosclerotic disease;
* creating a local registry (based on European CARDS percutaneous interventional registries) which also includes renal, metabolic and vascular data;
* reporting long-term follow-up data on major cardiac adverse events (MACE) in the study group.

DETAILED DESCRIPTION:
Gathered data:

* descriptive general demographic data;
* previous pathologies (ischemic heart disease, peripheral arterial disease, stroke, heart failure, previous percutaneous coronary interventions, coronary artery bypass grafting - CABG, known renal disease), cardiovascular risk factors (age, weight, height, abdominal perimeter, body mass index, smoking, sedentariness, diabetes, hypertension, dyslipidaemia);
* routine biological data and specific non-genetic biomarkers;
* information regarding primary PCI (less than 12 hours of ischemic symptoms): coronarographic details, type of used stent, periprocedural specific complications, final TIMI - thrombolysis in myocardial infarction - flow);
* echocardiography at admission (LVEF);
* metabolic data (obtained from body composition monitoring) - body water, body fat tissue;
* renal arteries angiographic details (two independent operators evaluate stenosis based on a predefined scale);
* renal dimensions;
* measurement of arterial stiffness through Sphigmocore pulsed-wave-velocity (24 hrs post-procedural, 2 velocities: carotid - femoral and carotid - radial);
* heart rate variability;
* in-hospital and one month follow-up MACE;

ELIGIBILITY:
Inclusion Criteria:

* adults with AMI (<12h) diagnostic confirmed;
* included in the Romanian National Programme of Primary Percutaneous Revascularisation (for who the Guidelines recommend primary PCI);

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * inclusion criteria: study population consists of all consecutive patients admitted with AMI (<12h) diagnostic confirmed;
  * included in the Romanian National Programme of Primary Percutaneous Revascularisation (for who the Guidelines recommend primary PCI);
  * have read and signed standard informed consent for angiography in AMI;
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
renal artery stenosis incidence | 2 years
  assessment of in renal artery stenosis incidence consecutive AMI patients included in the Romanian National Programme of Primary Percutaneous Revascularisation;

SECONDARY OUTCOMES:
cardio-renal-metabolic profile in patients with renal atherosclerotic disease; | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Burlacu, MD, Principal Investigator — University of Medicine and Pharmacy "Gr T Popa" Iasi
Locations (1):
- Cardiology Departament "IBCV" Hospital, Iași, Romania

REFERENCES:
- [Derived] Burlacu A, Siriopol D, Voroneanu L, Nistor I, Hogas S, Nicolae A, Nedelciuc I, Tinica G, Covic A. Atherosclerotic Renal Artery Stenosis Prevalence and Correlations in Acute Myocardial Infarction Patients Undergoing Primary Percutaneous Coronary Interventions: Data From Nonrandomized Single-Center Study (REN-ACS)-A Single Center, Prospective, Observational Study. J Am Heart Assoc. 2015 Oct 12;4(10):e002379. doi: 10.1161/JAHA.115.002379. PMID 26459932